CLINICAL TRIAL: NCT06497881
Title: Monitoring Post Stroke Upper-Limb Movement in The Wild
Brief Title: Upper Limb Movement Quality Following Stroke
Status: Recruiting | Type: Observational
Sponsor: Adi Negev-Nahalat Eran (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Sponsor
Other Study IDs: NegevLab_2024_1
Record Dates: First submitted 2024-07-01; First posted 2024-07-12 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stroke: Persons after a stroke. See inclusion/exclusion.
- Controls: Healthy persons. See inclusion/exclusion.

SUMMARY:
The aim of this study is to monitor the daily upper limb movement of persons with stroke, and to relate these quantities to measures of recovery and impairment.

DETAILED DESCRIPTION:
This study is part of The Natural History of Stroke Recovery project. In this study the investigators plan to develop, test and validate an algorithm and software for using Inertial Measuring Units (IMUs) to monitor upper limb daily movement. Then, investigators plan to use this system to monitor such activity in stroke patients.

Investigators also plan to develop, test and validate an algorithm and software to test proprioception acuity based on muscle synergy during active and passive movement. Muscle synergy will be determined based on muscles' electrical activity, as measured using surface electromyography (EMG).

Investigators will then test the relation between daily movements of the upper limb in stroke patients, and their recovery/impairment levels, including proprioception acuity.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Independent in all activities of daily living before the stroke.
* In- and out-patients at Adi-Negev Nahalat-Eran rehabilitation center.
* Medically stable
* Able to provide informed consent.

Exclusion Criteria:

* The presence of any degenerative neurological condition, neuropathy, myopathy or Polio that are not secondary to stroke, excluding diabetic related changes.
* Traumatic brain injury and/or extra-cerebral hemorrhage.
* Significant psychiatric condition, including alcoholism and drug abuse.
* Any severe orthopedic condition (such as amputation or severe pain that limits activity) or chronic pain syndrome.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons with stroke and healthy adults.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Hand movements-count | One or two occasions over 1-6 hours each.
  The number of hand movements (count)
Hand movements-duration | One or two occasions over 1-6 hours each.
  The total and average (per hour) time the hands moved, over the tested period. Measured in minutes.
Active joint range | One or two occasions over 1-6 hours each.
  Maximum, minimum, and mean range of motion of the joints during daily activity. Measured in degrees/radians.
Wrist distance | One or two occasions over 1-6 hours each.
  The maximum, average and total distance of the wrist from the body during movements. Measured in cm.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | One occasions during the first month following recruitment.
  Fugl-Meyer Assessment:
  Motor score of the upper limb is on a 0-66 scale. High score is better.
Action Research Arm Test (ARAT) | One occasions during the first month following recruitment.
  Action Research Arm Test Score is on a 0-57 scale. High score is better.
Proprioception-1 | One occasions during the first month following recruitment.
  The difference between joint angles in an angle matching task. E.g., matching the shoulder angle of a passively moved arm with the contralateral arm. Angles include both anatomical angles and elevation angles. Measured in degrees/radians.
Proprioception-2 | One occasions during the first month following recruitment.
  Parameters of the correlation (regression) between EMG signals during active and passive movement. Including the constant (in mV), slope (arbitrary units) and R^2 (arbitrary units).
Proprioception-3 | One occasions during the first month following recruitment.
  Delay between hand movement initiation observed kinematical (acceleration) and kinetically (EMG signal). Measured in msec.
Joint range of motion | One or two occasions over 1-6 hours each.
  Maximum and minimum joints range of motion (active and passive). Measured in degrees/radians.
Synergies | One or two occasions over 1-6 hours each.
  Parameters of the correlation (regression) between the kinematic signals of the different upper extremity segments. Including the slope (arbitrary units) and R^2 (arbitrary units).
Angular velocity. | One or two occasions over 1-6 hours each.
  Maximum and average angular velocity of the joints during daily activity. Measured in degrees/radians per second
Movement volume | One or two occasions over 1-6 hours each.
  Volume occupied by the limb segments calculated using the 3D location of the joints. Measured in cm^3.
Whole body movement time | One or two occasions over 1-6 hours each.
  The total and average (per hour) time of movements of the whole body. Measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Lior Smuelof, PhD, Principal Investigator — Ben-Gurion University of the Negev; Yogev Koren, PhD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Adi-Negev Nahalat Eran, Ofakim, Israel

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Will be available with publication of results, indefinitely.
Access Criteria: Open access.